CLINICAL TRIAL: NCT07301008
Title: Rimegepant as Preemptive Treatment for Predictable Trigger-Induced Migraine in Adult Patients in the US
Acronym: RIM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008797
Record Dates: First submitted 2025-10-20; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Migraine; Trigger Induced Migraine
Keywords: Trigger- induced migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rimegepant 75 MG (Experimental)
  Interventions: Drug: Rimegepant 75 MG

INTERVENTIONS:
Drug: Rimegepant 75 MG — The interventional product is rimegepant ODT 75 mg. Rimegepant 75mg ODT will be given 2 hours prior to a trigger exposure for exercise, alcohol (less than one drink per day for woman and less than two drinks per day for men), air travel that lasts no more than 12 hours, sexual activity, fasting that lasts no more than 24 hours rimegepant will be dosed 2 hours prior to trigger exposure. For weekend or let down headache and changes in sleep pattern, rimegepant will be dosed the night before. The maximum dose in a 24-hour period is 75mg.

SUMMARY:
Single-center, open label, prospective study conducted at Medstar Georgetown Headache Center. Men and woman ≥ 18 years old that are diagnosed with migraine with or without aura for at least 1 year, who report a reliable migraine trigger. Acceptable triggers for the study will include exercise, alcohol (less than one drink per day for woman and less than two drinks per day for men), air travel that lasts no more than 12 hours, sexual activity, fasting that lasts no more than 24 hours, stress or stress let-down headache.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 1 year history of episodic migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders-3 (ICHD-3)
* Men and women ≥ 18 years old .
* Average of 2-8 migraine attacks of moderate or severe intensity per month within the last 3 months prior to the screening visit
* Headache/migraine onset before age 50 years
* Migraine attacks, on average, lasting 4-72 hours if untreated
* At least 48 hours between migraine attacks
* Ability to distinguish migraine attacks from tension or cluster headaches
* Particpants on SOC treatment should be on stable regimen for at least 3 months prior to enrollment and should not change their regimen during the course of the study
* Participant may have been on treatment with Botox or mAbs for the last 6 months
* Participants experience migraine ≥75% of the time following exposure to a trigger during the run-in period. Acceptable triggers include exercise, alcohol ( less than one drink per day for woman and less than two drinks per day for men), air travel that lasts no more than 12 hours, sexual activity, fasting that lasts no more than 24 hours, stress or weekend/ let-down

Exclusion Criteria:

* Using gepants as preventive treatment (atogepant once daily (QD) or rimegepant every other day (EOD)), or using zavegepant or ubrogepant as an acute treatment
* History of use of narcotic or barbiturate containing medications, including opioids (e.g., morphine, codeine, oxycodone, and hydrocodone) on ≥5 days per month on a regular basis for ≥3 months prior to screening
* Current evidence of uncontrolled, unstable, or recently diagnosed cardiovascular disease, uncontrolled hypertension, or uncontrolled diabetes.
* Current diagnosis of major depressive disorder requiring treatment with atypical antipsychotics, schizophrenia, bipolar disorder, or borderline personality disorder.
* Women must not be pregnant, lactating or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of preemptive treatments with rimegepant in which migraine with a moderate to severe headache intensity | 24 hour post dose
  Percentage of preemptive treatments with rimegepant in which migraine with a moderate to severe headache intensity occurs within 24 hours

SECONDARY OUTCOMES:
Percentage of preemptive treatments with rimegepant | 24 hour, 48 hour post dose
  Percentage of preemptive treatments with rimegepant in which migraine occurs within 24 hours
  * Percentage of preemptive treatments with rimegepant that require rescue medication within 24 hours
  * Percentage of preemptive treatments with rimegepant that result in acute medication use within 48 hours of treatment
Patient satisfaction with preemptive treatment with rimegepant | At the end of the study completion( 2 month after enrollment)
  Patient satisfaction with preemptive rimegepant treatment will be assessed in the case report form using a Likert scale
The effect of preemptive treatment with rimegepant on Patient Global Impression of Change (PGIC) | At the end of study completion( 2 months after enrollement)
  The effect of preemptive treatment with rimegepant on Patient Global Impression of Change (PGIC) using a graded scale of 1-7.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ailani, MD, Principal Investigator — MedStar's Georgetown University Hospital
Locations (1):
- MedStar Health: Neurology at McLean, McLean, Virginia, United States

IPD SHARING:
Plan to Share IPD: No